CLINICAL TRIAL: NCT01050218
Title: A 9-Month Open-Label Extension Study of the Long-Term Safety of DVS SR in Outpatients With Pain Associated With Diabetic Peripheral Neuropathy
Brief Title: Study Evaluating the Long-Term Safety of Desvenlafaxine Succinate Sustained-Release (DVS SR) in Subjects With Pain Associated With Diabetic Peripheral Neuropathy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Business reasons
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3151A5-325
Record Dates: First submitted 2010-01-13; First posted 2010-01-15 (Estimated); Results first posted 2010-05-11 (Estimated); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Diabetic Neuropathy, Painful
Keywords: Diabetic Peripheral Neuropathy
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DVS SR Open Label (Other): Daily dose of 100mg or 200mg at the investigators discretion. Subjects already randomized at a dose of 400mg may continue at that dose level.
  Interventions: Drug: Desvenlafaxine Succinate Sustained-Release (DVS SR)

INTERVENTIONS:
Drug: Desvenlafaxine Succinate Sustained-Release (DVS SR)
  Other Names: DVS SR

SUMMARY:
The purpose of the study is to learn if long-term treatment with DVS SR is safe for treating the pain and other symptoms associated with diabetic peripheral neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients who have completed double-blind treatment in study 322 (NCT01050218) for DPN. Subjects must have completed all scheduled evaluations, with no major protocol violations and no events that, in the opinion of the investigator, would preclude the subject's entry into the long-term open-label study.
* Women of childbearing potential must have a negative serum pregnancy test on day 91 of the short-term study. A woman of childbearing potential is one who is biologically capable of becoming pregnant. "Biologically capable" includes women who are using contraceptives or whose sexual partners are either sterile or using contraceptives. Sexually active women participating in the study who are biologically capable of becoming pregnant must use a medically acceptable form of contraception during the study and for at least 15 days after the last dose of test article. Medically acceptable forms of contraception include oral contraceptives, transdermal, injectable, or implantable methods, intrauterine devices, or properly used double-barrier contraception, eg, condom plus diaphragm.

Exclusion Criteria:

* Presence of any new and/or clinically important medical condition that might compromise subject safety (including, but not limited to, significant changes in glycemic control).
* Pregnancy, lactation, or plans to become pregnant during the study.
* Use of prohibited treatments.
* Meets any of the exclusion criteria listed for study 322 (NCT01050218).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2006-07; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer

REFERENCES:
- [Derived] Allen R, Sharma U, Barlas S. Clinical experience with desvenlafaxine in treatment of pain associated with diabetic peripheral neuropathy. J Pain Res. 2014 Jun 23;7:339-51. doi: 10.2147/JPR.S55682. eCollection 2014. PMID 25018648

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited in the United States from July 2006 to September 2008.
Pre-assignment Details: Outpatients must have completed double-blind treatment and all scheduled evaluations in study 3151A5-322 (NCT00283842), with no major protocol violations and no events that, in the opinion of the investigator, would have precluded the subject's entry into the long-term open-label study.
Period: Overall Study
Arm/Group | DVS SR Open Label
Started | 237
Completed | 142
Not Completed | 95
Not completed — Adverse Event | 37
Not completed — Lack of Efficacy | 8
Not completed — Protocol Violation | 3
Not completed — Withdrawal by Subject | 18
Not completed — Discontinued by sponsor | 18
Not completed — Compliance | 2
Not completed — Failed to return | 7
Not completed — Serious Adverse Event | 1
Not completed — Family emergency | 1

BASELINE CHARACTERISTICS:
Arm/Group | DVS SR Open Label
Number analyzed (Participants) | 237
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.84 (8.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64
  Male | 173

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Pain Score on the Numeric Rating Scale (NRS).
Description: The primary efficacy variable was the pain severity score measured on an 11 point NRS on which 0=no pain and 10=worst possible pain. The primary efficacy evaluation was the change from baseline in mean pain score on the NRS.
Time Frame: Baseline and 9 months
Population: The efficacy population was the intent-to-treat (ITT). This included all randomized subjects who had a baseline primary efficacy evaluation, had taken at least 1 dose of test article, and had at least 1 primary efficacy evaluation (ie, at least 1 NRS daily pain score) after the first dose of test article. No participants met that criterion.
Arm/Group | DVS SR Open Label
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | DVS SR Open Label
Serious Adverse Events (participants affected / at risk) | 26/237
Other Adverse Events (participants affected / at risk) | 199/237
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DVS SR Open Label (N=237)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 3
Diastolic dysfunction (Cardiac disorders) | 1
Abdominal hernia (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Erosive oesophagitis (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 2
Asthenia (General disorders) | 1
Chest pain (General disorders) | 3
Oedema peripheral (General disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Cellulitis (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Localised infection (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Blood glucose fluctuation (Investigations) | 1
Blood glucose increased (Investigations) | 1
Blood pressure increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Haemorrhage intracranial (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Status epilepticus (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Mental status changes (Psychiatric disorders) | 2
Nephrolithiasis (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Ovarian mass (Reproductive system and breast disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Iliac artery stenosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DVS SR Open Label (N=237)
Ear and labyrinth disorders general (Ear and labyrinth disorders) | 12
Eye disorders general (Eye disorders) | 13
Diarrhoea (Gastrointestinal disorders) | 12
Dry mouth (Gastrointestinal disorders) | 15
Nausea (Gastrointestinal disorders) | 23
Vomiting (Gastrointestinal disorders) | 16
Fatigue (General disorders) | 13
Nasopharyngitis (Infections and infestations) | 19
Upper respiratory tract infection (Infections and infestations) | 24
Injury, poisoning and procedural complications general (Injury, poisoning and procedural complications) | 46
Investigations general (Investigations) | 38
Metabolism and nutrition disorders general (Metabolism and nutrition disorders) | 20
Arthralgia (Musculoskeletal and connective tissue disorders) | 14
Back pain (Musculoskeletal and connective tissue disorders) | 12
Muscle spasms (Musculoskeletal and connective tissue disorders) | 13
Dizziness (Nervous system disorders) | 39
Headache (Nervous system disorders) | 18
Psychiatric disorders general (Psychiatric disorders) | 35
Renal and urinary disorders general (Renal and urinary disorders) | 28
Reproductive system and breast disorders general (Reproductive system and breast disorders) | 13
Respiratory, thoracic and mediastinal disorders general (Respiratory, thoracic and mediastinal disorders) | 26
Skin and subcutaneous tissue disorders general (Skin and subcutaneous tissue disorders) | 37
Hypertension (Vascular disorders) | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs agreed to allow the sponsor 60 days to review and require changes to presentations or publications but only to protect confidential information and intellectual property, and for the sponsor to file a patent application, as applicable. The PIs also agreed for data to be presented first as a joint, multi-center publication.